# The efficacy of probiotics to reduce antepartum group B streptococcus colonization

# NCT03696953

Study protocol &

Statistical analysis plan 06-14-2018

Principle Investigator
Lisa Hanson PhD, CNM, FACNM, FAAN
Klein Professor
Marquette University,
College of Nursing,
Milwaukee, WI 53201-1881

# **Funding**

This research protocol and statistical analysis plan was supported by Eunice Kennedy Shriver National Institute of Child Health and Human Development of the National Institutes of Health under award number R21HD095320

#### Method

**Design.** The purpose of this Phase 2 placebo-controlled, double blind, randomized controlled trial (RCT) is to determine the efficacy of once daily ingestion of Florajen3 by healthy low-risk pregnant women from 28 weeks gestation until the time of labor to (a) reduce the proportion of women with GBS colonization and thus (b) reduce the number of women who receive IAP. We expect this intervention to alter the vaginal and rectal microbiota by (c) increasing *Lactobacillus* colony counts, (d) decreasing GBS colony counts, and (e) reducing GI symptoms.

Sample Size and Power Estimates. A provider group within the proposed study setting reported a 29.4% prevalence of GBS positive women among the 316 who gave birth in 2016. Therefore, we expect a 30% GBS prevalence in the placebo group compared to the probiotic group. To determine the effect size of the intervention, a sample of 80 women will be required to test the difference in proportions of GBS colonization and IAP between groups (hypotheses 1a and 1d). Hypotheses are unidirectional. With the sample size of 80 and setting alpha = 5%, one tailed test, 80% power estimate, and confounding variables (yogurt ingestion, vaginal cleansing practices, and sexual activity) accounting for multiple R-square = 0.1, we will be able to reject the null hypothesis for an effect size of Odds Ratio (OR) = 0.17 for the logistic regression to compare the proportion of GBS positives between groups. When comparing the colony counts (GBS and Lactobacillus) and GI symptoms (hypotheses 1b, 1c and 2), the same sample size = 80, power = 80%, alpha = 5%, one tailed test; we can reject the null hypothesis for a Cohen d = 0.56. This is a medium effect size, indicating that we can detect a difference between groups equivalent to 0.56 standard deviations. However, if the effect of the treatment is smaller we will be able to identify it, but not reject the null hypothesis of being equal to 0. This information is important for design of a full scale efficacy trial of the probiotic intervention. In our published preliminary study, 15 we found an overall dropout rate of 23%, but 30% in the probiotic group. For the proposed study, we chose a conservative 30% dropout rate to assure that the sample size can be fully achieved within the study timeline. Therefore, a total sample of 116 will be targeted for enrollment. Hypotheses 1b, 1c, and 2 will be tested by doing a multiple group comparison of the change in colony count for GBS and Lactobacillus, and the GI symptom inventory (M-SODA-9) scores [Section 2.3.1.8.e].

**Recruitment**. A sample of 116 women who meet the inclusion criteria, low-risk, healthy and pregnant,  $26 \pm 2$  weeks gestation, 18 years of age, will be recruited from a population of central city maternity care recipients who see either certified nurse-midwives or physicians at the prenatal clinics of Aurora Sinai Medical Center (ASMC) in Milwaukee, Wisconsin. Approximately 200 new prenatal patients are seen monthly. **Inclusion and exclusion criteria are detailed in Table 1.** 

Table 1. Study Inclusion and Exclusion Criteria

## **Inclusion Criteria**

Healthy adult (≥ 18 years of age) pregnant women who are 28±2 weeks gestation at enrollment [calculated from the first day of Last Normal Menstrual Period (LNMP) and/or ultrasound (US)]

With: No obstetric complication\* (e.g., pre-eclampsia, gestational diabetes, multiple gestation)

No fetal complication (e.g., birth defect, intrauterine growth restriction)

No medical complication (e.g., hypertension, diabetes mellitus)

Who do not currently ingest an over-the-counter probiotic supplement (not including yogurt)

Who can both speak and read English

Who regularly attend prenatal care appointments (defined as not > 1 prior missed appointment during this pregnancy)

## **Exclusion Criteria**

Pregnant women who have a history of GBS bacteriuria during the current pregnancy or have previously given birth to a GBS affected child

Women who are planning an elective repeat cesarean birth

<sup>\*</sup>Multigravidas with uncomplicated GBS colonization in a prior pregnancy will be eligible for participation in the study.

All participants regardless of group assignment will receive usual prenatal care. To facilitate recruitment, posters will be displayed in the waiting areas and in each prenatal examination room, and recruitment brochures will be available. The Study Coordinator (SC) will work with the clinic receptionist staff to identify women at 26 ± 2 weeks gestation on the day of their visit to the clinic. Participants will begin the study at 28 ± 2 weeks gestation. Once identified and introduced to the study by the SC, potential participants will be provided with a copy of the informed consent document. If she expresses an interest in the study, she will provide her name, due date, birth date, and phone number, as well as permission to be screened for study participation. The SC will conduct a prenatal chart review for study inclusion and exclusion criteria for each interested woman by completing the Prenatal Eligibility Screening Form (PESF)The SC will call the woman, thank her for her interest, and indicate whether she meets the study eligibility criteria. For those eligible and willing, the SC will arrange to meet the potential participant in the clinic just before her regularly scheduled prenatal visit at 28 ± 2 weeks gestation. Upon meeting, the SC will explain the study, review the informed consent (IC) document, and answer all questions, to complete IC procedures. The same setting and recruitment procedures were used for the team's preliminary study. 18 During the IC, participants will be apprised that they will begin taking oral study capsules once daily from 28 ± 2 weeks until labor. Participation is completed at 2 months postbirth. Intervention. Floraien3 is a combination probiotic with a once daily recommended dose. Each commercial batch of Florajen3 undergoes rigorous testing for potency, purity, and dose. Potency is maintained for 14 months when refrigerated. Subjects in the control group will take a daily placebo capsule of rice maltodextrin, identical in appearance, taste, and smell to the probiotic capsules. American Lifeline will ship the bulk probiotic and placebo products to the Aurora Investigational Drug Service (IDS) for the study.

Randomization Procedures, Preparation, and Allocation of Study Bottles. IDS consultants will randomize and prepare the study probiotic and placebo capsules, independent of Dr. Hanson and other study personnel. A simple randomization computer program will be used by the IDS consultants to generate the random number sequence used to randomly assign study participant numbers to receive either the probiotic or placebo capsules. The IDS staff will fill 58 bottles (each containing 112 probiotic pills) and 58 bottles (each containing 112 placebo pills) and label them in a manner that is blind to group assignment, indicating study numbers assigned from 1-116. The original list identifying the allocation and relationship to study number will be kept locked in the IDS, unavailable to Dr. Hanson or other study personnel until study completion, when unblinding will occur. Each study bottle will be covered with a MEMS cap (electronic cap counter) and placed in the refrigerator in the Aurora Sinai Medical Center Inpatient Pharmacy (ASMCIP). When the SC enrolls participants, retrieval of the prepared study bottles from the ASMCIP will occur with distribution of the specific participant's bottle that corresponds to the assigned study number.

**Intervention Initiation and Duration**. The **rationale** for third trimester (28 ± 2 weeks gestation) initiation of the probiotic intervention is based on the findings of our review of the scientific literature on antenatal probiotics. In 23 of the 31 RCTs included in our integrative review, the intervention was initiated in the third trimester without any adverse maternal, fetal, or neonatal outcomes. The intervention will be continued until labor to maintain microbiota effects (probiotic group) at the critical time for newborns. All participants will be instructed to keep the study bottle refrigerated and to take one capsule per day until they are in labor. We found no rationale to recommend "catch up" dosing if participants miss a capsule. Participants will return study bottles with any remaining unused capsules to SC at 1-2 days post birth.

Adherence. Adherence<sup>58</sup> will be measured in three ways: (a) A MEMS™ AARDEX™ electronic cap counter<sup>59</sup> will be placed on each numbered study bottle. Each opening of the bottle cap is recorded by an electronic chip that is linked to the SC's computer. (b) When bottles are returned during the post birth hospital stay, the remaining capsules will be counted to verify the MEMS cap count. (c) The qualitative 16S rRNA targeted sequencing method and PCR performed on vaginal and rectal swabs will recover probiotic bacteria contained in Florajen3. Two approaches designed to encourage participants' daily adherence are: (a) Each participant will receive a daily text message reminder<sup>60</sup> to take her study capsule. The participant will choose the timing of the daily text message. If the participant cannot receive text messages, she will be offered a refrigerator alarm. <sup>61,62</sup> (b) At prenatal and study visits participants will be reminded to take capsules daily.

**Procedure and Timing.** Table 2 contains a summary of data collection, variables, measures, and timing. Following IC, the SC will sequentially distribute the prelabeled, randomly numbered bottles of study capsules, as noted above. The SC will maintain a list of the participant names, linking them to the assigned study

numbers, in an encrypted computer file, accessible only to the PI and the SC. The PI, co-investigators, SC, prenatal providers, and participants will be blind to group assignment. Data will be collected at five time points: T1 baseline (28 ± 2 weeks), T2 (36 ± 2 weeks), T3 (1-2 days post birth, before hospital discharge), T4 (2 weeks post birth phone call), and T5 (2 months post birth follow-up phone call). Measures and documentation tools appear in Appendices A through G. At each study visit, participants will be asked about any potential adverse events. Immediately following IC, participants will have their first study visit at 28 ± 2 weeks gestation (T1), during which baseline data will be collected and they will receive instructions to take one capsule by mouth daily until the time of birth. Also at T1 (28 ± 2 weeks), the participant will be seen by her prenatal provider, who will facilitate collection of the baseline study samples. Participants will be asked to collect their own vaginal and rectal swabs with assistance, but have the option of provider collection. This minimally invasive testing does not require a speculum exam. Self-collected swabs yield similar colonization measures compared to provider-collected, but may be more acceptable to women. 63,64 Each participant will also complete three brief questionnaires at T1. Vaginal and rectal swabs and 2 questionnaires will be collected at T2 (36 ± 2 weeks). At the end of T2, participants will receive a \$25 gift card. At T3, the SC will visit every participant on the postpartum hospital unit to administer two brief questionnaires, retrieve the study bottle with MEMS cap, and give a \$75 gift card. The SC will analyze the MEMS cap data, count and record the capsules remaining in the bottle, and conduct a chart review. At T4 and T5, the SC will text message the participants to indicate that she/he will be phoning the next business day. The following day, a phone call will be made to the participant to elicit any maternal and child health events (e.g., illness, antibiotics, or hospital readmission). At T5, the SC will also retrieve health records for the participant and her infant to examine them for the same maternal or child health events.

Table 2. Summary of Study Data Collection, Variables, Measures, and Timing

| Outcome Variables | Study Data Collection | T1 | T2 | T3 | T4 | T5 |
|---|---|---|---|---|---|---|
| | SC will document data from all measures on the Summary | 28 ± 2 | 36 ± 2 | 1-2 days | 2 | 2 |
| | Data Collection Form (SDCF; Appendix B). | weeks | weeks | post- | weeks | months |
| | See Appendixes A-G for data collection forms for all | baseline | prenatal | birth | post- | post- |
| | procedures. | visit | visit | | birth | birth |
| | Procedures | | | | | |
| Qualitative GBS | Vaginal to rectal GBS swab. Collected at prenatal visit and | Not | X | Not | | |
| Colonization (+ or -) | sends to hospital lab, results found in record | indicated | | indicated | | |
| Quantitative GBS Colony | Separate vaginal and rectal GBS swabs. Collected at | X | X | | | |
| Counts | prenatal visit and SC send to Dr. Safdar's lab | | | | | |
| Quantitative Lactobacillus | Separate vaginal and rectal Lactobacillus swabs. Collected | X | X | | | |
| Colony Counts | at prenatal visit and SC mailed to Dr. Safdar's lab | | | | | |
| Intervention Adherence | Vaginal and rectal swabs collected at prenatal visit | | X | | | |
| | (presence of probiotic species verifies adherence) | | | | | |
| | 2. MEMS™AARDEX™ wireless electronic cap counter <sup>58,59</sup> | | | Х | | |
| | 3. Final Pill Count | | | Х | | |
| Maternal GI Symptoms | M-SODA-9 <sup>65,66</sup> GI symptom scale (completed by subject) | Х | Х | Х | | |
| IAP | IAP doses based on qualitative GBS result; also SC | | | Х | | |
| | records prenatal antibiotic exposures from medical record | | | | | |
| Demographics | Demographic characteristics Questionnaire | Χ | | | | |
| Questionnaire for Women | Questionnaire on diet containing yogurt, sexual practices, | Χ | Х | X | | |
| | vaginal cleaning practices (completed by study subject) | | | | | |
| Maternal-Infant Postbirth | SC interviews mother for maternal and infant health events | L | L | X | | L |
| Health | and potential adverse events; documents | <b></b> | | Х | TC | TC, HR |
| Adverse Events (AE) | Prenatal providers and SC solicit AE and document. | | Х | Х | TC | TC, HR |

Abbreviations: X = in-person study visit; TC = telephone call; HR = health record review.

- a. **Qualitative GBS Colonization.** Consistent with the CDC guidelines, between 35-37 weeks gestation (T2), the subject (or provider) will obtain a vaginal to rectal swab for GBS colonization to determine the need for IAP. [NOTE: In 2019, the guidelines changed and the prenatal GBS screens were collected at 36 weeks gestation.] The analysis of this swab will be done at the hospital laboratory and the result is reported as positive or negative for GBS. This swab will be done after the study swabs to prevent contamination of either site.
- b. **Quantitative GBS Colony Counts.** GBS colony counts, from separate vaginal and rectal swabs collected before the qualitative swabs, will be measured by Dr. Safdar's lab for this study, using CDC-recommended procedures to identify the number of GBS CFUs per swab (T1 & T2).
  - c. Quantitative Lactobacillus Colony Counts. The swabs of vaginal and rectal sites will be analyzed to

identify the actual number of Lactobacilli in each area, counted as CFUs per swab (T1 &T2).

- d. Intervention Adherence Measures
- d.1. **PCR** and **16s** rRNA **Targeted Sequencing**. Vaginal and rectal swabs for PCR and 16s rRNA targeted sequencing will be collected (T2) by the participant or her provider and sent to Dr. Safdar's lab for analysis to detect the presence of the probiotic strains contained in the probiotic intervention group, verifying adherence.
- d.2. **MEMS Caps.** Each opening of the MEMS<sup>™</sup> AARDEX<sup>™</sup> wireless electronic cap counters<sup>58,59</sup> will be recorded electronically with a software link to a study computer accessible to the SC and Dr. Hanson.
  - d.3. **Pill Counts.** The MEMS cap counts will be verified by the pill count when the bottle is returned.
- e. **Maternal GI Symptoms.** Because currently available GI quality of life scales focus on specific pathologies, we adapted the previously validated 7-item, non-pain symptom scale of the Severity of Dyspepsia Assessment (SODA)<sup>65</sup> (Cronbach's  $\alpha$  = 0.9) to operationalize this variable. For use during pregnancy, the symptoms of "diarrhea" and "constipation" were added, resulting in a 9-item scale. Participants rate the severity of each symptom over the past week on a 6-point Likert scale, ranging from 0 = *no problem, not present* to 5 = *very severe problem, markedly influences daily activities and/or requires rest.* The score on the 9 items is summed to arrive at a GI symptom score ranging 0-45. Our **Ante-Partum Gastrointestinal Symptom Inventory (AP-GI-SA)** was validated in a pilot study with a sample of 45 healthy pregnant women. <sup>66</sup> We found Cronbach's  $\alpha$  = 0.84, test-retest reliability, stability, and content and face validity (T1, T2, and T3).
- f. IAP. If GBS-positive, the number and type of IAP doses will be recorded by SC on the **Summary Data Collection Form (SDCF).** Additional prenatal and intrapartum antibiotic exposures for participants and infants will be recorded on this form by the SC as potential cofounding variables.
  - g. Potentially cofounding variables
  - g.1. Participants will complete the brief **Demographic Questionnaire (DQ)** at T1 only.
- g.2. Participants will complete the **Questionnaire for Women (Q4W)** at T1-T3 visits. To improve the reliability of subject recall, the Q4W asks for a report of the past week's ingestion of yogurt, vaginal cleansing practices, and sexual activity. The Q4W was used by the co-investigators in our preliminary study.<sup>18</sup>
- h. **Maternal-Infant Postpartum Health Events.** The SC will interview the participant for a history of postpartum health events for herself or the infant (T4 and T5) and document appropriately on two forms:
  - h.1. Maternal health events, recorded on Maternal Peripartal Health Check (MPHC).
  - h.2. Infant health events, recorded on Infant Health and Wellness Form (IHWF).
- i. **Adverse Events.** All providers and study personnel will solicit information about potential adverse events (AE) at each study visit (T2 through T5). Participants will be asked to report any suspected side effects or AE at any point in between study visits to their providers, who will then notify the PI, and follow the protocol established in the Human Subjects Section. AE will be recorded on **Q4W** (T2, T3), **MPHC and IHWF** (T4-T5). **Data Management.** Database and entry screens for this project will be developed using Epidata. To minimize errors, data will be double-entered and checked for invalid codes, values that are out of range, invalid dates, and skip patterns. All data will be verified against the original forms and imported to Epidata for analysis. **Descriptive Analyses.** Means, standard deviations or frequency distributions will be reported for all variables. We will test for differences in demographic characteristics of two groups (Florajen3 and placebo), including confounding variables such as sexual activity, vaginal hygiene practices, yogurt ingestion, and prenatal antibiotic use. Chi-square and independent *t* tests will be used to compare mode of birth, gestational age at birth, and birth weight and length, to assess equivalence of groups. Chi-square, Fischer's exact tests, and Wilcoxon methods will be used to test for difference among binary and categorical variables.

**Plan for Missing Data**. To estimate the overall treatment effect for the entire sample, an "intention to treat" analysis will be conducted, using our above likelihood-based analysis method for repeated measures, including data on all subjects who were randomized to study groups, thus allowing us to use all available data, rather than delete participants with missing values from the analysis of treatment effects. <sup>67,68</sup> Pattern mixture modeling <sup>69</sup> will be used to understand the effects of protocol compliance. Thus, treatment effectiveness during the full intended duration of the protocol can be compared with the effectiveness of treatments while participants are compliant with them. <sup>70</sup>

**Binary Outcomes Analyses: Aim 1.** Using an intention-to treat approach, subjects will not be dropped from any preliminary analysis due to varying degrees of adherence with their group-specific therapy. The main hypothesis, 1a, along with hypothesis 1d, assess differences in proportions, and will be analyzed using a generalized linear model (GLM).<sup>71,72</sup> Those response variables that are dichotomous (binomial distribution) will be analyzed using the logit link to assess the proportional difference in GBS-colonized women (hypothesis 1a)

and the proportion of women requiring IAP (hypotheses 1d). GLM allows us to include confounding variables in the same model providing an effect size measure for the treatment and confounding variables, the odds ratio (OR), which has direct interpretation as the odds difference of testing GBS positive.

**Continuous Outcomes Analyses: Aims 1 and 2.** A secondary analysis of research aims 1 and 2 will be conducted using a Gaussian distribution-based multilevel generalized linear mixed model to assess group differences in GBS (hypothesis 1 b) and *Lactobacillus* (hypothesis 1c) colony count changes from 28 weeks to 35-37 weeks, <sup>73</sup> with time points (T1-T2) nested within subjects. Group differences can be estimated for both initial time point and slope. The treatment is expected to show a meaningful difference to the slope of colony count change. Confounding variables will be included as time-invariant covariates. Parameters that appear to be meaningless will be excluded, using log-likelihood (deviance) model comparison with a direct interpretation as the colony count slope difference between groups, which can be transformed into a standardized difference (Cohen's *d*).

**Confirmatory Factor Analysis: Aim 2.** The GI symptom scale will be analyzed using a confirmatory factor analysis (CFA)<sup>74</sup> using R Version 3.3.1 or later.<sup>75</sup> With a multiple group CFA, we will compare the GI symptoms construct mean and variance between the placebo and treatment groups (hypothesis 2). Confounding variables will be included as covariates, estimating their effects for each group separately.

## References

- Verani JR, McGee L, Schrag SJ. Prevention of perinatal group B streptococcal disease. Revised guidelines from CDC, 2010. MMWR Morb Mortal Wkly Rep. 2010; 59(RR-10);1-32. https://www.cdc.gov/mmwr/preview/mmwrhtml/rr5910a1.htm
- 2. Centers for Disease Control and Prevention (CDC). Prevention of perinatal group B streptococcal disease. Revised guidelines from CDC. MMWR Morb Mortal Wkly Rep. 2002; 51(RR-11):1-22.
- 3. Ohlsson A, Shah VS. Intrapartum antibiotics for known maternal Group B streptococcal colonization. Cochrane Database Syst Rev. 2014(3). doi:10.1002/14651858.CD007467.
- 4. McKeever TM, Lewis SA, Smith C, Collins J, Heatlie H, Frischer M, Hubbard R. Early exposure to infections and antibiotics and the incidence of allergic disease: a birth cohort study with the West Midlands General Practice Research Database. J Allergy Clin Immunol. 2002;109(1):43-50.
- 5. de Vrese M. Health benefits of probiotics and prebiotics in women. Menopause Int. 2009;15:35.
- 6. Bizzarro MJ, Dembry L-M, Baltimore RS, Gallagher PG. Changing patterns in neonatal Escherichia coli sepsis and ampicillin resistance in the era of intrapartum antibiotic prophylaxis. Pediatrics. 2008;121:689-696.
- 7. Vangay P, Ward T, Gerber JS, Knights D. Antibiotics, pediatric dysbiosis, and disease. Cell Host Microbe. 2015;17(5):553-564.
- 8. Bedford Russell AR, Murch SH. Could peripartum antibiotics have delayed health consequences for the infant? BJOG. 2006;113:758-765.
- 9. Ecker KL, Donohue PK, Kim KS, Shepard JA, Aucott SW. The impact of group B streptococcus prophylaxis on late-onset neonatal infections. J Perinatol. 2013;33(3):206-211.
- 10. Aloisio I, Mazzola G, Corvaglia LT, Tonti G, Faldella G, Biavati B, et al. Influence of intrapartum antibiotic prophylaxis against group B streptococcus on the early newborn gut composition and evaluation of the anti-streptococcus activity of *Bifidobacterium* strains. Appl Microbiol Biot. 2014;98(13):6051-6060.
- 11. Keski-Nisula L, Kyynarainen H-R, Karkkainene, U, Karhukorpi J, Heinanen S, Pekkanen J. Maternal intrapartum antibiotics and deceased vertical transmission of *Lactobacillus* to neonates during birth. Acta Paediatr. 2013;102:480-485.
- 12. Buckler B, Bell J, Sams R, Cagle W, Bell SA, Allen C, Sutherland D, Bhatia J. Unnecessary workup of asymptomatic neonates in the era of Group B Streptococcus prophylaxis. Infect Dis Obstet Gynecol. 2010; Article ID 369654, 3 pages.
- 13. Hanson L, VandeVusse L. Group B streptococcus intrapartum prophylaxis guidelines adherence: a perinatal risk management issue. J Perinat Neonatal Nurs. 2010;24(2):100-103.
- 14. White House. National Strategy for Combating Antibiotic-resistant Bacteria. Washington, DC; 2014 (September). Accessed January 20, 2016. Available from: https://www.whitehouse.gov/sites/default/files/docs/carb\_national\_strategy.pdf
- 15. Allen SJ. Dietary supplementation with Lactobacilli and Bifidobacteria is well tolerated and not associated with adverse events during late pregnancy and early infancy. J Nutr. 2010;140(3):483-488.
- 16. VandeVusse L, Hanson L, Safdar N. Perinatal outcomes of prenatal probiotic and prebiotic administration: an integrative review. J Perinat Neonat Nurs. 2013; 27(4):288-301.
- 17. Ephraim E, Schultz RD, Duster M, Warrack S, Spiegel C, Safdar N. In-vitro evaluation of antagonistic effects of the probiotics *Lactobacillus* rhamnosus HN001 and Florajen3 against Group B streptococci. Int J Probiotics Prebiotics. 2012;7(3/4):113-120.
- 18. Hanson L, VandeVusse L, Duster M, Warrack S, Safdar N. Feasibility of oral prenatal probiotics against maternal Group B Streptococcus vaginal and rectal colonization. J Obstet Gynecol Neonatal Nurs. 2014;43:294-304.
- 19. Gregory KE. Microbiome aspects of perinatal and neonatal health. J Perinat Neonatal Nursing. 2011;25(2):158-162.
- 20. Hickmann ME, Rench MA, Ferrieri P, Baker CJ. Changing epidemiology of group B streptococcal colonization. Pediatrics. 1999; 104:203-209.
- 21. Cunningham FG, Leveno KJ, Bloom SL, Hauth JC, Rouce DJ, Spong CY. Infectious diseases: bacterial infections. In: Williams Obstetrics. 23rd ed. New York, NY: McGraw Hill; 2010:1220-1223.
- 22. Reid G, Dols J, Miller W. Targeting the vaginal microbiota with probiotics as a means to counteract infections. Curr Opin Clin Nutr Metab Care. 2009;12:583-587.

- 23. Ehrstrom S, Daroczy K, Rylander E, <u>Samuelsson C</u>, <u>Johannesson U</u>, <u>Anzén B</u>, et al. Lactic acid bacteria colonization and clinical outcome after probiotic supplementation in conventionally treated bacterial vaginosis and vulvovaginal candidiasis. <u>Microbes Infect</u>. 2010;12(10):691-699. doi:10.1016/j.micinf.2010.04.010. Epub 2010 May 28.
- 24. Hemmerling A, Harrison W, Schroeder A, Park J, Korn A, Shiboski S, et al. Phase 2a study assessing colonization efficiency, safety, and acceptability of *Lactobacillus* crispatus CTV-05 in women with bacterial vaginosis. Sex Transm Dis. 2010;37(12):745-750.
- 25. Stapleton AE, Au-Yeung M, Hooton TM, <u>Fredricks DN</u>, <u>Roberts PL</u>, <u>Czaja CA</u>, et al. Randomized, placebo-controlled Phase 2 trial of a *Lactobacillus* crispatus probiotic given intravaginally for the prevention of recurrent urinary tract infection. <u>Clin Infect Dis.</u> 2011;52(10):1212-1217. doi:10.1093/cid/cir183. Epub 2011 Apr 14.
- 26. Ronnqvist PDJ, Forsgren-Brusk UB, Hakansson EEG. Lactobacilli in the female genital tract in relation to other genital microbes and vaginal pH. Acta Obstet Gynecol. 2006;85:726-735.
- 27. Moghaddam MN. Recto-vaginal colonization of Group B Streptococcus in pregnant women referred to a hospital in Iran and its effect on *Lactobacillus* normal flora. <u>J Biol Sci</u>. 2010;10(2):166-169.
- 28. Berthier, A., Senthiles, L, Hamou L, Renoult-Litzer D, Marret S, Marpeau L. Antibiotics at term. Questions about five allergic accidents. Gynecol Obstet Fertil. 2007;35:464-72.
- 29. Jao M-S, Cheng P-J, Shaw S-W, Soong Y-K. Anaphylaxis to Cefazolin during labor secondary to prophylaxis for Group B Streptococcus: a case report. J Reprod Med. 2006;51:655-658.
- 30. Unger JA, Whimbey E, Gravett MG, Eschenbach DA. <u>The emergence of Clostridium difficile infection among peripartum women: a case-control study of a C. difficile outbreak on an obstetrical service.</u> Infect Dis Obstet Gynecol 2011; Article ID 267249, 8 pages.
- 31. Turrentine MA, Ramirez MM, Mastrobattista JM. Cost-effectiveness of universal prophylaxis in pregnancy with prior Group B Streptococci colonization. Infect Dis Obstet Gynecol. 2009; Article ID 934698, 11 pages.
- 32. Isaacs D, Unnatural selection: reducing antibiotic resistance in neonatal units. Arch Dis Child Fetal Neonatal Ed. 2006;91:F72-F74.
- 33. Glasgow TS, Young PC, Wallin J, Kwok C, Stoddard G, Firth S, Samore M, Byington CL. Association of intrapartum antibiotic exposure and late-onset serious bacterial infections in infants. Pediatrics. 2005;116:696-702.
- 34. Edwards MS. Issues of antimicrobial resistance in Group B Streptococcus in the era of intrapartum antibiotic prophylaxis. Semin Pediatr Infect Dis J. 2006;17:149-152.
- 35. Koenig JM, Keenan WJ. Group B Streptococcus and early-onset sepsis in the era of maternal prophylaxis. Pediatr Clin N Am. 2009;56:689-708.
- 36. Chohan L, Hollier LM, Bishop K, Kilpatrick CC. Patterns of antibiotic resistance among Group B Streptococcus isolates: 2001-2004. Infect Dis Obstet Gynecol. 2006; Article ID 57492, 4 pages.
- 37. Edwards RK, Clark P, Sistrom CL, Duff P. Intrapartum antibiotic prophylaxis 1: relative effects of recommended antibiotics on gram-negative pathogens. Obstet Gynecol. 2002;100:534-539.
- 38. Gritz EC, Bhandari V. The human neonatal gut microbiome: a brief review. Front Pediatr. 2015;3:Article 17, 12 pages. http://dx.doi.org/10.3389/fped.2015.00017
- 39. National Institutes of Health, National Human Genome Research Institute. Frequently asked questions about clinical research: What are clinical trial "phases?" Accessed May 30, 2017. Available from: https://www.genome.gov/10000771/.
- 40. Joint FAO/WHO Working Group Report on Drafting Guidelines for the Evaluation of Probiotics in Food. Guidelines for the evaluation of probiotics in food. London, Ontario, Canada: Author; April-May 2002. Accessed July 4, 2013. Available from: <a href="http://www.fda.gov/ohrms/dockets/dockets/95s0316/95s-0316-rpt0282-tab-03-ref-19-joint-faowho-vol219.pdf">http://www.fda.gov/ohrms/dockets/dockets/95s0316/95s-0316-rpt0282-tab-03-ref-19-joint-faowho-vol219.pdf</a>
- 41. Reid JNS, Bisanz JE, Monachese M, Burton JP, Reid G. The rationale for probiotics improving reproductive health and pregnancy outcome. Am J Reprod Immunol. 2013;69(6):558-566.
- 42. Food and Agriculture Organization of the United Nations & World Health Organization (FAO/WHO). Report on Joint FAO/WHO Expert Consultation on Evaluation of Health and Nutritional Properties of Probiotics in Food including Powder Milk with Live Lactic Acid Bacteria. Cordoba, Argentina: Author; 2001. Accessed July 4, 2013. Available from: <a href="http://www.who.int/foodsafety/publications/fs\_management/en/probiotics.pdf">http://www.who.int/foodsafety/publications/fs\_management/en/probiotics.pdf</a>

- 43. Elias J, Bozzo P, Einarson A. Are probiotics safe for use during pregnancy and lactation? Can Fam Physician. 2011;57:299-301.
- 44. Dugoua J-J, Machado M, Zhu X, Chen X, Koren G, Einarson TR. Probiotic safety in pregnancy: a systematic review and meta-analysis of randomized controlled trials of *Lactobacillus*, *Bifidobacterium*, and Saccharomyces spp. J Obstet Gynaecol Can. 2009;31(6):542-552.
- 45. Naaktgeboren CA. Effects of maternal probiotic exposure during pregnancy and lactation on the mother and infant. Int J Probiotics Prebiotics. 2010;5(3):113-124.
- 46. Myhre R, Brantsaeter AL, Myking S, Gjessing HK, Sengpiel V, Meltzer HM, et al. Intake of probiotic food and risk of spontaneous preterm delivery. Am J Clin Nutr. 2011;93:15 1-157.
- 47. Brantsaeter AL, Myhre R, Haugen M, Myking S, Sengpiel V, Magnus P, et al. Intake of probiotic food and risk of preeclampsia in primiparous women: The Norwegian mother and child cohort study. Am J Epidemiol. 2011;174(7):807-815.
- 48. Kim LS, Hilli L, Orlowski J, Kupperman JL, Baral M, Waters RF. Efficacy of probiotics and nutrients in functional gastrointestinal disorders: a preliminary clinical trial. Dig Dis Sci. 2006;51:2134-2144.
- 49. Lindsay KL, Kennelly M, Culliton M, Smith T, Maguire OC, Shanahan F, et al. Probiotics in obese pregnancy do not reduce maternal fasting glucose: a double-blind, placebo-controlled, randomized trial (Probiotics in Pregnancy Study). Am J Clin Nutr. 2014;99:1432-1439. doi:10.3945/ajcn.113.079723. Epub 2014 Mar 19.
- 50. Oostdam N, van Poppel MN, Wouters MG, van Mechelen W. Interventions for preventing gestational diabetes mellitus: a systematic review and meta-analysis. J Womens Health (Larchmt). 2011;20(10):1551-1563. 1:10.1089/jwh.2010.2703. Epub 2011 Aug 12. Review. PMID: 21838525
- 51. Azad, MB, Coneys JG, Kozyrskyj AL, Field CJ, Ramsey CD, Becker AB, et al. Probiotic supplementation during pregnancy or infancy for the prevention of asthma and wheeze: systematic review and meta-analysis. BMJ. 2013;347:f6741.
- 52. Doege K, Grajecki D, Zyriax B-C, Detinkina E, zu Eulenburg C, Buhling K J. Impact of materal supplementation with probiotics during pregnancy on atopic eczema in childhood: a meta-analysis. <u>Br J Nutr.</u> 2012;107:1-6.
- 53. Lee J, Seto D, Bielory L. Meta-analysis of clinical trials of probiotics for prevention and treatment of pediatric atopic dermatitis. *J Allergy Clin Immunol*. 2008;121:116-121.
- 54. Panduru M, Panduru NM, Salavastru CM, Tiplica GS. Probiotics and primary prevention of atopic dermatitis: a meta-analysis of randomized controlled studies. *J Eur Acad Dermatol Venereol*. 2015;29:232-42.
- 55. Pelucchi C, Chatenoud L, Turati F, Galeone C, Moja L, Bach J-F, La Vecchia C. Probiotics supplementation during pregnancy or infancy for the prevention of atopic dermatitis: a meta-analysis. *Epidemiology*. 2012;23(3):402-414.
- 56. Laitinen K, Poussa T, Isolauri E. Nutrition, Allergy, Mucosal Immunology and Intestinal Microbiota Group. Probiotics and dietary counseling contribute to glucose regulation during and after pregnancy: a randomised controlled trial. Br J Nutr. 2009;101:1679–1687.
- 57. Hanson L, VandeVusse L, Abad C, Safdar N. Probiotics for treatment and prevention of urogenital infections in women: a systematic review. J Midwifery Womens Health; 2016, 61:339-355.
- 58. Finigan J, Naylor K, Paggiosi MA, Peel NF, Eastell R. Adherence to raloxifene therapy: assessment methods and relationship with efficacy. Osteoporos Int. 2013;37(7):790-794.
- 59. Robiner WN, Flaherty N, Fossum TA, Nevins TE. Desirability and feasibility of wireless electronic monitoring of medications in clinical trials. Transl Behav Med. 2015;5(3):285–293. http://doi.org/10.1007/s13142-015-0316-1
- 60. Thakkar J, Kurup R, Laba T-L, Santo K, Thiagalingam A, Rodgers A, et al. Mobile telephone text messaging for medication adherence in chronic disease: a meta-analysis. JAMA Internal Med. 2016;176(3):340-349.
- 61. Haynes RB, Ackloo E, Sahota N, McDonald HP, Yao X. Interventions for enhancing medication adherence. Cochrane Database Syst Rev. 2008(2):CD000011.
- 62. Frick PA, Lavreys L, Mandaliya K, Kreiss JK. Impact of an alarm device on medication compliance in women in Mombasa, Kenya. Int J STD AIDS. 2001;12(5):329-333.

- 63. Arya A, Cryan B, O'Sullivan K, Greene RA, Higgins JR. Self-collected versus health professional-collected genital swabs to identify the prevalence of group B Streptococcus: a comparison of patient preference and efficacy. Eur J Obstet Gynecol Reprod Biol. 2008;139(1):43–45. doi:10.1016/j.ejogrb.2007.12.005
- 64. Mercer BM, Taylor MC, Fricke JL, Baselski VS, Sibai BM. The accuracy and patient preference for self-collected group B Streptococcus cultures. Am J Obstet Gynecol. 1995;173(4):1325–1328. doi:10.1016/0002–9378(95)91380–7
- 65. Rabeneck L, Cook KF, Wristers K, Souchek J, Menke T, Wray NP. SODA (severity of dyspepsia assessment): a new effective outcome measure for dyspepsia-related health. J Clin Epidemiol. 2001;54:755-765.
- 66. Hanson L, VandeVusse L, Garnier-Villarreal M, McCarthy D, Jerofke-Owen T, Malloy E, Paquette H. Validity and Reliability of the Antepartum Gastrointestinal Symptom Assessment Instrument. J Obstet Gynecol Neonatal Nurs. 2020 May;49(3):305-314. doi: 10.1016/j.jogn.2020.02.006. Epub 2020 Apr 6. PMID: 32272088.
- 67. Chakraborty H, Gu, H. (2009). A mixed model approach for intent-to-treat analysis in longitudinal clinical trials with missing values. RTI Press publication No. MR-0009-0903. Research Triangle Park, NC: RTI International. Accessed June 10, 2015. Available from: http://www.rti.org/rtipress.
- 68. Nich C, Carroll KM. (2002). 'Intention-to-treat' meets 'missing data': Implications of alternate strategies for analyzing clinical trials data. Drug Alcohol Depend. 2002;68(2):121-130.
- 69. Hedeker D, Gibbons RD. (1997). Application of random-effects pattern-mixture models for missing data in longitudinal studies. Psychol Meth. 1997;2:64-78.
- 70. Buuren S. Flexible imputation of missing data. Boca Raton, FL: CRC Press; 2012.
- 71. Brown H, Prescott R. Applied mixed models in medicine. 2nd ed. Chichester, West Sussex, England: Wiley & Sons; 2006.
- 72. Liu H, Wu T. Sample size calculation and power analysis of time-averaged difference. J Mod App Stat Meth. 2005;4(2):434-445.
- 73. Gelman A, Hill J. Analytical methods for social research: data analysis using regression and multilevel/hierarchical models. New York: Cambridge University Press; 2006.
- 74. Little TD. Longitudinal structural equation modeling: methodology in the social sciences. New York: Guilfors Press; 2013.
- 75. R core team. R: a language and environment for statistical computing. Vienna, Austria: R Foundation for Statistical Computing; 2016. Accessed April 15, 2017. Available from: <a href="https://www.R-project.org/">https://www.R-project.org/</a>.